CLINICAL TRIAL: NCT04793074
Title: Transforming Nanoparticle Dressing For Management of Chronic Venous Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EBRN080321
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Chronic Venous Hypertension With Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transforming nanoparticle dressing (Experimental): Patients in the treatment group (n=30) had transforming nanoparticle dressing
  Interventions: Combination Product: Transforming nanoparticle dressing
- Conventional compression dressing (Active Comparator): The control group (n=30) received conventional compression dressing.
  Interventions: Combination Product: Conventional compression dressing

INTERVENTIONS:
Combination Product: Transforming nanoparticle dressing — Transforming nanoparticle dressing
  Arms: Transforming nanoparticle dressing
Combination Product: Conventional compression dressing — Conventional compression dressing
  Arms: Conventional compression dressing

SUMMARY:
The present randomized controlled study aims to evaluate the role of transforming nanoparticle dressing n management of chronic venous ulcers.

DETAILED DESCRIPTION:
The present randomized controlled study was conducted at Helwan University Hospitals, Cairo, Egypt. The study protocol was approved by the local ethical committee and all patients gave informed consent before enrollment.

The study included 60 patients with CVU. Patients were diagnosed on the basis of clinical findings and vascular Doppler ultrasonography. Exclusion criteria were associated infection and associated ulcers of other etiologies. Patients randomization was achieved using computer generated numbers and sealed envelope technique. Randomization and patients' allocation to the study interventions was performed by an independent researcher who wasn't aware of the study interventions and outcome.

Upon recruitment, patients were subjected to careful history taking, thorough clinical examination, standard laboratory investigations and vascular ultrasound examination. The recorded parameters included demographic data (age, sex and body mass index), associated morbidities, duration and size of CVU and history of previous interventions.

After randomization, patients in the treatment group (n=30) had transforming nanoparticle dressing while the control group (n=30) received conventional compression dressing. Before applications of both dressings, the wound area was thoroughly cleaned. In the treatment group, the dressing powder was applied as a thin layer to the ulcer surface. Any excess powder surrounding the ulcer area was removed. In both groups, a secondary protective gauze dressing was applied. Patients were follow up at weekly intervals until complete healing occurs.

The primary end-point in the present study is the time to complete healing. The secondary end-point the rate of healing (percent of reduction in ulcer area).

ELIGIBILITY:
Inclusion Criteria:

* Chronic venous ulcers.

Exclusion Criteria:

- Associated infection and associated ulcers of other etiologies.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Time to complete healing (weeks) | 16 weeks
  The primary end-point in the present study is the time to complete healing of ulcers

CONTACTS AND LOCATIONS:
Overall Officials: Barakat Abdelreheem, Principal Investigator — Helwan University
Locations (1):
- Helwan University, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahmood BA, ElSayed EH, Abd Elghany SM, Elnaggar DF, Youssef HAA, Abdelmaksoud SM. A New Powder Dressing for Management of Chronic Venous Ulcers. Dermatol Surg. 2023 Jul 1;49(7):664-668. doi: 10.1097/DSS.0000000000003812. Epub 2023 Apr 25. PMID 37134230